CLINICAL TRIAL: NCT01216345
Title: Cetuximab Plus Gemcitabine-Oxaliplatin (GEMOX) in Patients With Unresectable Advanced or Metastatic Biliary Tract Cancer: a Phase II Study
Brief Title: Cetuximab + Gemox in Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Association of Research on the Biology of Liver Tumors (Other)
Responsible Party: Association of Research on the Biology of Liver Tumors
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CCC 01
Record Dates: First submitted 2010-10-04; First posted 2010-10-07 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2010-10

CONDITIONS: Unresectable; Locally Advanced; Metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Cetuximab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetuximab + Gemcitabine + Oxaliplatin — Cetuximab 500mg/m2, iv every two weeks Gemcitabine 1000mg/m2, iv every two weeks Oxaliplatin 100mg/m2, iv every two weeks
  Other Names: Erbitux; GEMOX

SUMMARY:
The aim of this prospective single-centre phase II study is to investigate the therapeutic efficacy and safety of cetuximab in combination with Gemcitabine and Oxaliplatin (GEMOX) in the palliative first line treatment of biliary tract cancer (BTC) patients.

DETAILED DESCRIPTION:
Primary Objective(s) The primary objective of the study is to evaluate the best overall response of cetuximab in combination with gemcitabine and oxaliplatin (GEMOX) as first line treatment in patients with advanced or metastatic biliary tract cancer.

Secondary Objectives

The secondary objectives of this study are as follows:

* toxicity
* secondary resection rate
* progression-free survival (PFS)
* overall survival (OS)

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically proven unresectable advanced or metastatic biliary tract cancer (including intrahepatic and extrahepatic CC and gallbladder cancer)
* age ≥ 18 years
* ECOG performance status ≤ 2
* bidimensionally measurable disease per RECIST criteria
* no prior chemotherapy or targeted therapy for advanced disease
* adequate bone marrow reserve (neutrophil count > 1500 /µL, platelet count > 100,000 /µL)
* adequate renal function (serum creatinine ≤ 1.5 x the upper limit of normal)
* adequate hepatic function (serum bilirubin <2.5 x the upper limit of normal (ULN) and serum transaminase level of ≤ 5 x ULN)
* written informed consent

Exclusion Criteria:

* prior palliative treatment
* resectable disease
* brain metastases
* serious or uncontrolled concurrent medical illness
* pregnancy or nursing
* history of other malignancies with the exception of excised cervical or basal skin/squamous cell carcinoma
* peripheral neuropathy (grade > 1)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-10; Primary Completion 2008-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
best overall response (according to RECIST 1.0) | after an average of 2 months
  overall response rate (ORR) will be measured after each 4 cycles (average 2 months) of Cetuximab +GEMOX and the overall best response recorded

SECONDARY OUTCOMES:
Safety of the treatment combination | approximately 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- KH Rudolfstiftung, Vienna, Austria

REFERENCES:
- [Result] Gruenberger B, Schueller J, et al: K-ras status and response in patients with advanced or metastatic cholangiocarcinoma treated with cetuximab plus gemcitabine-oxaliplatin (GEMOX): a single center phase II study J Clin Oncol 27:15s, 2009 (suppl; abstr 4586)
- [Derived] Gruenberger B, Schueller J, Heubrandtner U, Wrba F, Tamandl D, Kaczirek K, Roka R, Freimann-Pircher S, Gruenberger T. Cetuximab, gemcitabine, and oxaliplatin in patients with unresectable advanced or metastatic biliary tract cancer: a phase 2 study. Lancet Oncol. 2010 Dec;11(12):1142-8. doi: 10.1016/S1470-2045(10)70247-3. Epub 2010 Nov 9. PMID 21071270